CLINICAL TRIAL: NCT02473237
Title: Efficacy and Acute Effects on Walked Distance froM basEline and Post Dose of indacateRol vs Tiotropium in Women With modeRAte to Severe COPD Secondary to Biomass Exposure: Open Label Crossover Clinical Trial
Brief Title: Efficacy in Walked Distance of Indacaterol vs Tiotropium in Women With COPD Secondary to Biomass (EMERALD)
Acronym: EMERAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Principal Investigator, Alejandra Ramirez Venegas, MD, National Institute of Respiratory Diseases, Mexico
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C 22-12
Record Dates: First submitted 2015-05-22; First posted 2015-06-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: COPD
Keywords: COPD; biomass
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- indacaterol (Experimental): Indacaterol 150 mcgr, one inhaled capsule, dose once time on visit one, with dry powder inhaler device.
  Interventions: Drug: indacaterol
- Tiotropium (Active Comparator): Tiotropium 18 mcgr, 1 inhaled capsule, dose once time a Day, with dry powder inhaler device.
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: indacaterol — Indacaterol, one inhales capsule, 150 mcgr, by dry powder dispositive
  Other Names: Onbrize
  Arms: indacaterol
Drug: Tiotropium — Tiotropium 18 mcgr, one inhaled capsule, by dry powder inhaler handihaler
  Other Names: Spiriva
  Arms: Tiotropium

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) secondary to biomass exposure constitutes a chronic respiratory condition frequently excluded from large clinical trials. Biomass exposure COPD have some histopathologic, clinical, radiological and functional differences with tobacco smoke COPD. However, until now, there are no evidence in this patients about the clinical response to bronchodilators routinely used in tobacco smoke COPD.

Primary objective: To compare changes in walked meters from baseline on six minute walking test (6MWT) to 23:45 hours after one dose of indacaterol vs tiotropium in patients with moderate to severe COPD secondary to biomass exposure.

Secondary objectives: To compare changes in pulmonary function (inspiratory capacity, Forced Expiratory Volume in first second (FEV1) milliliters, FEV1 "through") from baseline (-10 minutes) to 23:45 hours after one dose of indacaterol vs tiotropium in patients with moderate to severe COPD secondary to biomass exposure.

This will be an open label study, double blinded, cross over and conducted at specialized respiratory care center (National Institute of Respiratory Diseases), to compare the acute effects of ultra long acting bronchodilators used in tobacco smoke exposure COPD. Unicentric study.

Ethics Committee approbation: C 22-12

DETAILED DESCRIPTION:
Background: Until now, COPD secondary to biomass exposure is treated in similar way that COPD due to tobacco smoke. Unfortunately none of the clinical trial included patient with biomass exposure in their multicenter studies. COPD due to biomass exposure is very common in Mexico and in other sub-developed countries, and represent a high economy burden similar as the tobacco exposure. In Mexico, in a reference center of COPD (National Institute of Respiratory Disease) thirty percent of women who attended with COPD has only the antecedent to cook with biomass. These patients have a predominant airway component, rather than emphysema. These patients have chronic bronchitis as a main clinical picture and in consequence, more exacerbations. Additionally, they present more symptoms such as dyspnea, and as COPD secondary to tobacco exposure, the functional and inspiratory capacity are reduced. There are previous studies that described the acute effects of long acting bronchodilators like salmeterol on functional and inspiratory capacity. However, they were done in patients with COPD secondary to tobacco smoke and there are not studies done in patients with COPD secondary to biomass exposition. Indacaterol a novel long-acting bronchodilator provide 24 h bronchodilation on once-daily dosing with a fast onset of action. Assuming the conditions of patients with COPD secondary to biomass exposure (women, rural or suburban origin, etc.) it is necessary strategies that enhance the adherence. There is information about better adherence with the least frequency of a drug. Tiotropium provide 24 h bronchodilation on once-daily dosing with a slow onset of action, it was selected because it is widely used in the treatment of COPD and is the only drug of the therapeutic class (long acting antimuscarinic bronchodilator) available in the market.

Until now there is no international nor national reported experience with any bronchodilators in COPD secondary to biomass.

This will be the first clinical trial in the world that attempts to evaluate the acute effects (fast onset action) of those two long acting bronchodilators, in women with COPD secondary to biomass exposure. Besides, the results will help to highlight the need in the rest of the world to include these patients in the different multicenter studies.

Primary objective:

To compare changes in walked meters from baseline six minute walking test (6MWT) to 23:45 hours after one dose of Indacaterol (150µg) vs Tiotropium (18µg) in patients with moderate to severe COPD secondary to biomass exposure.

Secondary efficacy Objectives are:

1. To compare changes in Inspiratory Capacity (IC) from baseline (-10 minutes) to 30, 60, 240 minutes and 23:45 hours post dose of Indacaterol (150 µg) vs Tiotropium (18µg) in patients with with biomass smoke COPD.
2. To compare changes in FEV1 from baseline (-10 minutes) to 30, 60, 240 min and 23:45 hours post dose of Indacaterol (150 µg) vs Tiotropium (18µg) in patients with biomass smoke COPD.
3. To compare the 'trough' FEV1 (mean of values at 23 h 10 min and 23 h 45 min post-dose) after one dose of indacaterol vs tiotropium in patients with COPD secondary to biomass exposure.
4. To compare changes in dyspnea perception by using the Borg scale from baseline (-10 minutes) to 30, 60, 240 min and 23:45 hours post dose of Indacaterol (150 µg) vs Tiotropium (18 µg) in patients with COPD secondary to biomass exposure.
5. To compare the frequency of adverse events presented during the study, between indacaterol vs tiotropium arm.

Methodology:

This will be an open label study conducted at specialized respiratory care center (National Institute of Respiratory Diseases, Mexico) to compare the 24 hours response to two long acting bronchodilators (Indacaterol vs Tiotropium), after one inhaled dose.

The primary endpoint will be changes in walked meters (6MWT) from baseline to 30, 60, 120 and 240 minutes post dose of Indacaterol (150 µg) vs Tiotropium (18µg) in patients with moderate to severe COPD secondary to biomass exposure.

The key secondary endpoint will be the 'trough' FEV1 in milliliters (mean of values at 23 h 10 min and 23 h 45 min) post dose of Indacaterol (150 µg) vs Tiotropium (18 µg) in patients with moderate to severe COPD secondary to biomass exposure.

The "trough" FEV1 value which was based on the mean of two measurements taken 23 h 10 min and 23 h 45 min following the previous day's morning dose.

Other secondary endpoints will be:

* FEV1 (in milliliters) and Inspiratory Capacity (IC in milliliters) will be measured frpm baseline (-10 min) to 30, 60, 90, 120 and 240 minutes post bronchodilators.
* Dyspnea perception will be measured by the 10 points Borg scale, from baseline to 30, 60, 120 and 240 minutes post bronchodilators.

In all patients spirometry will be performed serially over 24 h postdose. The design implies a crossover treatment in order to avoid variability between subjects and guarantee the outcome measures.

There will be 40 intervention patients with 40 controls (crossover design). The study comprised a pre-screening visit, a 7-day screening period, and one day, 1-week treatment periods. At the baseline visit, eligible patients were randomized equally to one of two treatment sequences (A or B) to receive either indacaterol 150 µg once-daily or Tiotropium 18 µg once-daily, followed by the other bronchodilator (Tiotropium or Indacaterol) each of them via a single-dose dry powder inhaler (SDDPI). Each treatment period was separated by a washout period of 7 days.

Number of centers & patients: 1 center with 40 patients, sequentially exposed to the two option treatment and will be their own control. It was decided making a self control design with crossover treatment in order to avoid variability between subjects and guarantee the outcome measures.

Sample size justification:

The sample size was calculated considering a power of 80% and a alpha value of 0.05 and two tails. Taking the minimal clinical significance value for 6 minutes walking test of 54 meters and standard deviation of 95 meters (BODE study). Because of the design of the study the investigators expected minimal patient withdrawn (less than 10%).

Population:

It is known that COPD secondary to biomass exposure patients commonly have a frequent exacerbation phenotype compared with patients with COPD secondary to tobacco smoke, and the investigators also expect that this phenotype would have the major benefit of the therapy. That´s why there will be included COPD patients in groups B, C or D, according to GOLD update 2011.

Pharmacovigilance requirements:

All the Adverse Events (AE) would be reported following the procedure for Serious Adverse Events (SAEs) Report. In order to guarantee the safety of the patient, any AE occurring after patients began with the treatment of indacaterol.

All the recurrence, complications or progression of the original AE must be reported as follow up of the original event, no matter when it was presented. This report should be submitted during the first 24 hours after the treating physician receive the notification. Any AE that is not considered to be related to the previous reported AE, should be informed as a new event.

All SAEs shall be collected and registered in Serious Adverse Event Report Form.

Outcome measurements:

Primary:

Walked meters on six minute walking test.

Secondary:

inspiratory capacity and post bronchodilator measures changes from basal measures .

1. Changes from baseline in pulmonary function and inspiratory capacity.
2. Changes from baseline in the total score of the Borg scale for dyspnea measure.

ELIGIBILITY:
Inclusion Criteria:

1. Mexican patients at the COPD outpatient clinic
2. Age: >50
3. Female (female eligibility criteria are: Women in no fertile age who are non pregnant and committed to use effective contraception).
4. FEV1 less than 80% of predicted and risk of exacerbation (GOLD update 2011) B, C or D
5. Women with COPD diagnostic with biomass exposition (defined with an Hours/years index >200 hr/y).
6. Be Able to assist at the different visits during the study.
7. Be Able to performed the spirometry
8. Patients without contraindications to perform the six-minute walk test.
9. Informed consent signed.
10. No history of exacerbations in the last 6 weeks previous to the inclusion.
11. With amenorrhea history more than a year duration.

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Use of Methotrexate, gold salts, troleandomycin, cyclosporine, immunosuppressants,
3. History of uncontrolled renal disease, liver disease, uncontrolled cardiovascular disease, metabolic disease, neurologic disease, hematologic disease, oncologic disease, or autoimmune disease.
4. Any alteration in normal values of the following Laboratory test: liver test, PIE, Biochemistry tests.
5. History of asthma, bronchiectases, tuberculosis, recent respiratory tract infection, were hospitalized for a COPD exacerbation (6 weeks prior to visit 1), any significant pulmonary disease o cardiovascular abnormality
6. Patients that is under suspicion of having cancer.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
changes in walked meters on six minute walking test (6MWT) from baseline to 23:45 hours after one dose of indacaterol vs tiotropium in patients with moderate to severe COPD secondary to biomass exposure. | baseline, 30, 60, 240 and 23:45 hours post dose of indacaterol vs tiotropium

SECONDARY OUTCOMES:
changes in Inspiratory Capacity (IC) from baseline (-10 minutes) to 30, 60, 240 minutes and 23:45 hours post dose of Indacaterol (150 µg) vs Tiotropium (18µg) in patients with with biomass smoke COPD. | baseline, 30, 60, 240 and 23:45 hours post dose of indacaterol vs tiotropium
the 'trough' FEV1 (mean of values at 23 h 10 min and 23 h 45 min post-dose) after one dose of indacaterol vs tiotropium in patients with COPD secondary to biomass exposure. | 23:10 and 23:45 hours post dose of indacaterol vs tiotropium
changes in dyspnea perception by using the Borg scale from baseline (-10 minutes) to 30, 60, 240 min and 23:45 hours post dose of Indacaterol (150 µg) vs Tiotropium (18 µg) in patients with COPD secondary to biomass exposure. | baseline, 30, 60, 240 and 23:45 hours post dose of indacaterol vs tiotropium
the frequency of adverse events presented during the study, between indacaterol vs tiotropium arm | 4 weeks
  non serious adverse events; serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Ramírez-Venegas, M.Cs., Principal Investigator — Instituto Nacional de Enfermedades Respiratorias, "Ismael Cosío Villegas"
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, "Ismael Cosío Villegas", Mexico City, Mexico City, Mexico

REFERENCES:
- [Result] Perez-Padilla R, Regalado J, Vedal S, Pare P, Chapela R, Sansores R, Selman M. Exposure to biomass smoke and chronic airway disease in Mexican women. A case-control study. Am J Respir Crit Care Med. 1996 Sep;154(3 Pt 1):701-6. doi: 10.1164/ajrccm.154.3.8810608.
- [Result] Bruce N, Perez-Padilla R, Albalak R. Indoor air pollution in developing countries: a major environmental and public health challenge. Bull World Health Organ. 2000;78(9):1078-92. PMID 11019457
- [Result] Torres-Duque C, Maldonado D, Perez-Padilla R, Ezzati M, Viegi G; Forum of International Respiratory Studies (FIRS) Task Force on Health Effects of Biomass Exposure. Biomass fuels and respiratory diseases: a review of the evidence. Proc Am Thorac Soc. 2008 Jul 15;5(5):577-90. doi: 10.1513/pats.200707-100RP. PMID 18625750
- [Result] Regalado J, Perez-Padilla R, Sansores R, Paramo Ramirez JI, Brauer M, Pare P, Vedal S. The effect of biomass burning on respiratory symptoms and lung function in rural Mexican women. Am J Respir Crit Care Med. 2006 Oct 15;174(8):901-5. doi: 10.1164/rccm.200503-479OC. Epub 2006 Jun 23. PMID 16799080
- [Result] Caballero A, Torres-Duque CA, Jaramillo C, Bolivar F, Sanabria F, Osorio P, Orduz C, Guevara DP, Maldonado D. Prevalence of COPD in five Colombian cities situated at low, medium, and high altitude (PREPOCOL study). Chest. 2008 Feb;133(2):343-9. doi: 10.1378/chest.07-1361. Epub 2007 Oct 20. PMID 17951621
- [Result] Ramirez-Venegas A, Sansores RH, Perez-Padilla R, Regalado J, Velazquez A, Sanchez C, Mayar ME. Survival of patients with chronic obstructive pulmonary disease due to biomass smoke and tobacco. Am J Respir Crit Care Med. 2006 Feb 15;173(4):393-7. doi: 10.1164/rccm.200504-568OC. Epub 2005 Dec 1. PMID 16322646
- [Result] Aaron SD, Vandemheen KL, Fergusson D, Maltais F, Bourbeau J, Goldstein R, Balter M, O'Donnell D, McIvor A, Sharma S, Bishop G, Anthony J, Cowie R, Field S, Hirsch A, Hernandez P, Rivington R, Road J, Hoffstein V, Hodder R, Marciniuk D, McCormack D, Fox G, Cox G, Prins HB, Ford G, Bleskie D, Doucette S, Mayers I, Chapman K, Zamel N, FitzGerald M; Canadian Thoracic Society/Canadian Respiratory Clinical Research Consortium. Tiotropium in combination with placebo, salmeterol, or fluticasone-salmeterol for treatment of chronic obstructive pulmonary disease: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):545-55. doi: 10.7326/0003-4819-146-8-200704170-00152. Epub 2007 Feb 19. PMID 17310045